CLINICAL TRIAL: NCT04805957
Title: A Pilot Project to Validate Digital Bio-markers as a Tool to Measure Improvement in Core Symptoms of Autism During Sulforaphane Treatment.
Brief Title: Validation Digital Bio-markers During Sulforaphane Treatment.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Elizabeth B. Torres Ph.D., Associate Professor of Psychology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2019001854
Record Dates: First submitted 2020-07-09; First posted 2021-03-18 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Autism; Autism Spectrum Disorder; Autistic Disorder
Keywords: Sulforaphane
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: This is a 12 week open label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All subjects will receive 1.47umol/kg/day sulforaphane for 12 weeks. Pills are taken once a say with a meal.
  Interventions: Dietary Supplement: Sulforaphane

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Sulforaphane comes from eating certain cruciferous vegetables. In this case the pills are made from broccoli seeds.
  Other Names: Avmacol®

SUMMARY:
The purpose of the research is to determine if changes seen during sulforaphane treatment (a compound that comes from eating certain vegetables) can better be understood using digital biomarkers. These digital biomarkers are things like heart rate, muscle movement etc. and are measured using non-invasive devices (like a watch) and are aimed at complementing the traditional clinical scores already in use in current trials (e.g. Aberrant Behavior Checklist (ABC), Social Responsiveness Scale (SRS) and Ohio Autism Clinical Impressions Scale (OACIS)).

DETAILED DESCRIPTION:
This study is a pilot open label treatment trial with SF (sulforaphane) in 10 individuals that have completed with moderate to severe autism, age 13-30 years that have completed participation in ClinicalTrials.gov Identifier: NCT02677051. This study will measure digital biomarkers of the nervous systems. Digital biomarkers are obtained by using non-invasive wireless (wearable, like wearing a watch) biosensors that co-register in tandem multiple biorhythms self-generated by the person's nervous systems. These sensors gather a very large amount of data from measures such as EEG (electroencephalogram), EKG (electrocardiogram), kinematics and others. These measures are done at the same time as the clinical evaluations and so results can be compared. Because the data are based on the unique fingerprint-like signatures of the person's nervous systems, it is possible to ascertain the person's progression in response to treatment and compare it to baseline states. The project will also compare these self-emerging clusters between subjects, possibly identifying patterns that correlate with sub-phenotypes or with similarities in response to treatment. Changes in things such as natural behaviors, an individual's ability or desire to interact socially and ability or desire to communicate will alter the signature profiles from baseline. Since these changes are dynamic in nature, trends of the evolving patterns and separate changes that are a consequence of the treatment vs. changes that are part of the natural neurodevelopment can be detected. This may be a valuable tool in future studies of underlying etiology. The technology used to perform these measures and the software to analyze the data are evolving rapidly. Last, with the characterized signatures and possibly overlapping patterns generated in this and in other projects it is foreseeable that a clinically relevant tool for measures in autism will follow.

ELIGIBILITY:
Inclusion Criteria:

* Autistic disorder diagnosis.
* Age between 13-30 years.
* Male gender.
* Participated in clinical trial NCT02677051

Exclusion Criteria:

* Those that started or continued taking Avmacol® or similar broccoli extracts since leaving our double-blind study.
* Absence of a parent or legal guardian and consent,
* Those that can not or will not complete all visits and adherence to study regimen.
* Seizure within 2 years of screening,
* History of chronic kidney, liver or thyroid disease.
* Impaired renal function (serum creatinine> 1.2 mg/dl).
* Impaired hepatic function (> 2x upper limit of normal).
* Impaired thyroid function (TSH outside normal limits).
* Current infection or treatment with antibiotics.
* Chronic medical disorder (e.g., cardiovascular disease, stroke or diabetes) or major surgery within 3 months prior to enrollment.
* Less than 13 years or more than 30 years of age.
* Female gender.
* A diagnosis of autism spectrum disorder other than autistic disorder, for example, Asperger, PDD-NOS ( Pervasive Developmental Disorder-Not Otherwise Specified) etc.

Ages: 13 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist (ABC) | Baseline.
  Rating scale to measure severity aberrant behaviors
Aberrant Behavior Checklist (ABC) | Week 6.
  Rating scale to measure severity aberrant behaviors
Aberrant Behavior Checklist (ABC) | Week 12, end of treatment.
  Rating scale to measure severity aberrant behaviors
Aberrant Behavior Checklist (ABC) | Week 16.
  Rating scale to measure severity aberrant behaviors
Social Responsiveness Scale (SRS) | Baseline.
  Rating scale to measure social interaction.
Social Responsiveness Scale (SRS) | Week 6.
  Rating scale to measure social interaction.
Social Responsiveness Scale (SRS) | Week 12, end of treatment.
  Rating scale to measure social interaction.
Social Responsiveness Scale (SRS) | Week 16.
  Rating scale to measure social interaction.
Ohio Autism Clinical Global Impression Scale - Severity (OACIS-S, an autism specific version of the Clinical Global Impression, CGI) | Baseline.
  Rating scale to measure autism severity and changes in severity.
Ohio Autism Clinical Global Impression Scale - Severity (OACIS-S, an autism specific version of the Clinical Global Impression, CGI) | Week 6.
  Rating scale to measure autism severity and changes in severity.
Ohio Autism Clinical Global Impression Scale - Severity (OACIS-S, an autism specific version of the Clinical Global Impression, CGI) | Week 12, end of treatment.
  Rating scale to measure autism severity and changes in severity.
Ohio Autism Clinical Global Impression Scale - Severity (OACIS-S, an autism specific version of the Clinical Global Impression, CGI) | Week 16.
  Rating scale to measure autism severity and changes in severity.
Digital Biomarkers | Baseline.
  Non-invasive biosensor measurements of micro-movements.
Digital Biomarkers | Week 6.
  Non-invasive biosensor measurements of micro-movements.
Digital Biomarkers | Week 12, end of treatment.
  Non-invasive biosensor measurements of micro-movements.
Digital Biomarkers | Week 16.
  Non-invasive biosensor measurements of micro-movements.
EEG | Baseline
  Electroencephalogram (EEG) measures electrical activity of the brain.
EEG | Week 6.
  Electroencephalogram (EEG) measures electrical activity of the brain.
EEG | Week 12, end of treatment.
  Electroencephalogram (EEG) measures electrical activity of the brain.
EEG | Week 16.
  Electroencephalogram (EEG) measures electrical activity of the brain.
EKG | Baseline
  Electrocardiogram (ECG or EKG) measures electrical signals from the heart.
EKG | Week 6.
  Electrocardiogram (ECG or EKG) measures electrical signals from the heart.
EKG | Week 12, end of treatment.
  Electrocardiogram (ECG or EKG) measures electrical signals from the heart.
EKG | Week 16.
  Electrocardiogram (ECG or EKG) measures electrical signals from the heart.
Electrophysiological recordings. | Baseline
  Measurement of electrical activity in Tissue.
Electrophysiological recordings. | Week 6.
  Measurement of electrical activity in Tissue.
Electrophysiological recordings. | Week 12, end of treatment.
  Measurement of electrical activity in Tissue.
Electrophysiological recordings. | Week 16.
  Measurement of electrical activity in Tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers-RWJMS Department of Neurology, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh K, Connors SL, Macklin EA, Smith KD, Fahey JW, Talalay P, Zimmerman AW. Sulforaphane treatment of autism spectrum disorder (ASD). Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15550-5. doi: 10.1073/pnas.1416940111. Epub 2014 Oct 13. PMID 25313065
- [Background] Torres EB, Brincker M, Isenhower RW, Yanovich P, Stigler KA, Nurnberger JI, Metaxas DN, Jose JV. Autism: the micro-movement perspective. Front Integr Neurosci. 2013 Jul 24;7:32. doi: 10.3389/fnint.2013.00032. eCollection 2013. PMID 23898241
- [Background] Torres EB. Atypical signatures of motor variability found in an individual with ASD. Neurocase. 2013 Apr;19(2):150-65. doi: 10.1080/13554794.2011.654224. Epub 2012 May 16. PMID 22587379

DOCUMENTS (1):
  • Informed Consent Form (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT04805957/ICF_000.pdf